CLINICAL TRIAL: NCT04544176
Title: Determining the Risk of Developing Symptomatic SARS-COV2-19 Infection After Attending Hospital for Radiological Examinations: a Controlled Cohort Study
Brief Title: COVID-19 Risk From Attending Outpatient Radiology Appointments
Status: Completed | Type: Observational
Sponsor: Nottingham University Hospitals NHS Trust (Other)
Collaborators: University Hospital of Wales (Other)
Responsible Party: Sponsor
Other Study IDs: 20NS031
Record Dates: First submitted 2020-09-09; First posted 2020-09-10 (Actual); Last update posted 2021-02-12 (Actual); Status verified 2021-02

CONDITIONS: Covid19
Keywords: Radiology; Outpatient; Hospital
MeSH Terms: conditions — COVID-19 | interventions — Watchful Waiting

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Exposed Cohort: This group will include patients attending radiology outpatient appointments in 2020 in our period of interest from the peak of the first wave of the pandemic, who were subsequently tested for SARS-COV2 within 28-days of their attendance.
  Interventions: Other: Observational
- Unexposed Cohort: This group will form the control group and comprises all individuals who attended radiological appointments during the same period for each hospital in 2019 but not 2020.
  Interventions: Other: Observational

INTERVENTIONS:
Other: Observational — There will be no interventions in this study, it is purely observational using data already collected.

SUMMARY:
By using recent data on hospital attendance and COVID-19 laboratory tests, available within two NHS trusts in Nottingham and Cardiff we will enable the calculation of the risk of developing COVID-19 infection after attending an outpatient hospital appointment. This will assist in the restart planning when resuming face to face outpatient radiology appointment.

DETAILED DESCRIPTION:
Since March 2020, the novel coronavirus (COVID-19) pandemic has caused considerable disruption to the provision of routine healthcare in the UK. A key priority for healthcare providers when gaining control of COVID-19, is to restart the provision of urgent non-COVID care. There are several barriers including a reluctance for people to attend hospital appointments for fears of contracting COVID-19. Although SARS-COV2 infections have been reported to occur during hospital inpatient stay, the risk of acquiring SARS-COV2 during outpatient consultations or radiological investigations has not been reported.

In a pilot study at our hospitals during the pandemic, we have found radiology to reliably record in person attendance contrary to outpatient clinic appointments records that were contaminated by remote consultations. The investigators will calculate the incidence of infection in approximately 30,000 patients at Nottingham and 17,000 patients at Cardiff and calculate the risk of infection within 28 days of attending outpatient radiology appointments. Controls will use data on patients who attended the hospitals in 2019.

The study team will utilize the data held in the electronic systems of NUH and University Hospital of Wales to perform a cohort study which will comprise both an exposed cohort and unexposed cohort.

The exposed cohort will comprise patients who attended outpatient radiology appointments during (between 29/1/20 - 24/5/20) and whether they subsequently developed a positive or negative PCR test for Sars-CoV2 result within 28-days of their attendance. The unexposed cohort will work as a control group, comprising individuals who attended outpatient radiology appointments during the equivalent period in 2019.

All of this data will be retrospective, so will not require any additional data collection, nor will it interfere with routine clinical care. Pseudo-anonymised data will be transferred from University Hospital of Wales in Cardiff to Nottingham University Hospitals (NUH) Trust via a password-protected, encrypted spreadsheet, with original patient identifiers removed, and a unique code assigned, that only the researcher in Cardiff can use to trace back to the individual, this is so all the analysis can be performed at NUH by a Nottingham based statistician.

The study team consisting of clinicians, data analysts, epidemiologist and clinical researchers will analyse this information to quantify the risk of infection which will help inform the recovery plans and service provision during the restart of urgent and routine non-COVID care.

ELIGIBILITY:
Inclusion Criteria:

Exposed Cohort: outpatient radiology attendance at NUH between 29/1/20 - 24/5/20 or at University Hospital of Wales, Cardiff between 7/3/20 - 11/5/20.

Unexposed Cohort: outpatient attendance outpatient attendance at NUH between 29/1/19 - 24/5/19 or at University Hospital of Wales, Cardiff between 7/3/19 - 11/5/19.

Exclusion Criteria:

Patients who had an inpatient stay in the previous 28-days but excluding the 2 days prior to the SARS-COV2 test Radiological examinations that were part of an inpatient stay were not considered

Ages: 16 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: All individuals attending outpatient clinics will be included for analysis, this is anticipated this to be in excess of 30,000 patients at NUH and around 17,000 patients at Cardiff. To ensure a substantive number of patients are included for analysis and comparison across the UK, 2 large hospitals (Nottingham University Hospitals and Cardiff University Hospitals) will be participating in this study.
Sampling Method: Non-Probability Sample
Enrollment: 48000 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2020-06-30 (Actual); Study Completion 2021-01-01 (Actual)

PRIMARY OUTCOMES:
A microbiological diagnosis of COVID infection. | 6 months
  Information will be collected on patients who receive a positive or negative COVID-19 test.

CONTACTS AND LOCATIONS:
Overall Officials: Nikos Evangelou, FRCP, DPhil (Oxon), Principal Investigator — University of Nottingham
Locations (1):
- Nottingham University Hospitals, NHS Trust, Nottingham, Nottinghamshire, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided